CLINICAL TRIAL: NCT02939703
Title: Integrating Quantitative Energetics Determines the Microbiome's Contribution to Energy Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TRIMD FH 942699
Record Dates: First submitted 2016-09-16; First posted 2016-10-20 (Estimated); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Obesity
Keywords: Adipose tissue; calorimetry; energy expenditure; microbiome
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Western diet (Active Comparator): Participants will consume a control western diet prepared by our metabolic research kitchen for an outpatient period followed by an inpatient period.
  Interventions: Other: Diet
- Microbiome Enhancer diet (Experimental): Participants will consume an experimental microbiome enhancer diet prepared by our metabolic research kitchen for an outpatient period followed by an inpatient period
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Participants will consume either a Control Western Diet or a Microbiome Enhancer Diet.

SUMMARY:
We propose to study the role of the gut microbiome in the development of obesity, and whether we can change the microbiome's contribution to host energy balance through diet. We have created a novel model that explicitly links the effects of microorganisms on human energy balance and modeled weight change, and will use the power of metabolic ward studies to measure small changes in energy absorption, total daily energy expenditure, and/or food intake that affect long-term weight gain or loss. By integrating clinical measurements, bioreactor experiments, and mathematical modeling, we will be able to describe cause-and-effect mechanisms that will enable a quantification of the microbiota's contribution to weight gain and inspire future studies on the interactions of diet, the gut microbiome, and human physiology.

ELIGIBILITY:
Inclusion Criteria:

1. Able to communicate meaningfully with the investigator and legally competent to provide informed written consent
2. Age 18 - 45 years, inclusive
3. Weight stable (+/- 3 kg) during the 6 months prior to enrollment
4. BMI ≤ 30 kg/m2

Exclusion Criteria:

1. History or presence of cardiovascular disease (unstable angina, myocardial infarction or coronary revascularization within 6 months, clinically significant abnormalities on EKG, presence of cardiac pacemaker, implanted cardiac defibrillator)
2. History of type 1 or type 2 diabetes
3. Bleeding disorders
4. Acute or chronic infections
5. Hepatitis and/or cirrhosis
6. Severe asthma or chronic obstructive pulmonary disease
7. Renal insufficiency or nephritis
8. Thyroid dysfunction (suppressed TSH, elevated TSH if symptomatic, elevated thyroid stimulating hormone (TSH) if asymptomatic)
9. Uncontrolled hypertension (BP >160 mmHg systolic or >100 mmHg diastolic)
10. Prior bariatric surgery
11. Inflammatory bowel disease or malabsorption, swallowing disorders, suspected or known strictures, fistulas or physiological/mechanical GI obstruction, history of gastrointestinal surgery, Crohn's disease or diverticulitis
12. Participants with strict dietary concerns (e.g. vegetarian or kosher diet, multiple food allergies, or allergies to food we will provide them during the study)
13. Current use of polyethylene glycol (e.g. Dulcolax, Miralax, Gavilax)
14. Cancer within the last 3 years (except non-melanoma skin cancer or treated cervical carcinoma in situ)
15. History of depression within < 5 years from screening visit or which, in the opinion of a medical investigator, will impact the participant's ability to complete the study
16. History of eating disorders
17. Cushing's disease or syndrome
18. Untreated or inadequately controlled hypo- or hyperthyroidism
19. Active rheumatoid arthritis or other inflammatory rheumatic disorder
20. Pregnant or nursing females or females less than 6 months postpartum from the scheduled date of collection.
21. Tobacco use within the past 3 months
22. Metal implants (pace-maker, aneurysm clips) based on Investigator's judgment at Screening.
23. Unable to participate in MRI or MRS assessments due to physical limitations of equipment tolerances (e.g. MRI bore size) based on Investigator's judgment at Screening.
24. Unable to tolerate MRI/MRS imaging or claustrophobia.
25. Nickel allergy.
26. Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pretrial (screening) visit.
27. Intolerance to acetaminophen use.
28. History of regular alcohol consumption exceeding 7 drinks/week for female participants or 14 drinks/week for male participants (1 drink = 5 ounces [150 mL] of wine or12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
29. Anemia (hemoglobin <12 g/dl in men, <11 g/dl in women)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for the protocol is the within-participant difference in fecal energy (via chemical oxygen demand, COD) normalized to the total daily energy intake and to the non-metabolizable marker PEG [COD (kcal) / PEG (g)]. | Days 24-29 vs. Days 53-58
  Comparison within subject of control diet versus microbiome enhancer diet.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, MD, Principal Investigator — Study Principal Investigator; Rosa Krajmalnik-Brown, PhD, Principal Investigator — Study Principal Investigator at Arizona State University
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Igudesman D, Yu G, Dutta T, Carnero EA, Krajmalnik-Brown R, Smith SR, Corbin KD. Global Metabolite Profiling in Feces, Serum, and Urine Yields Insights into Energy Balance Phenotypes Induced by Diet-Driven Microbiome Remodeling. Am J Clin Nutr. 2025 Oct;122(4):1027-1041. doi: 10.1016/j.ajcnut.2025.08.003. Epub 2025 Aug 19. PMID 40835099
- [Derived] Corbin KD, Carnero EA, Dirks B, Igudesman D, Yi F, Marcus A, Davis TL, Pratley RE, Rittmann BE, Krajmalnik-Brown R, Smith SR. Host-diet-gut microbiome interactions influence human energy balance: a randomized clinical trial. Nat Commun. 2023 May 31;14(1):3161. doi: 10.1038/s41467-023-38778-x. PMID 37258525
- [Derived] Corbin KD, Krajmalnik-Brown R, Carnero EA, Bock C, Emerson R, Rittmann BE, Marcus AK, Davis T, Dirks B, Ilhan ZE, Champagne C, Smith SR. Integrative and quantitative bioenergetics: Design of a study to assess the impact of the gut microbiome on host energy balance. Contemp Clin Trials Commun. 2020 Aug 19;19:100646. doi: 10.1016/j.conctc.2020.100646. eCollection 2020 Sep. PMID 32875141
- See also: Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org/

DOCUMENTS (1):
  • Informed Consent Form (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT02939703/ICF_000.pdf